CLINICAL TRIAL: NCT03739840
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled, Parallel-Group Study to Evaluate the Efficacy and Safety of Padsevonil as Adjunctive Treatment of Focal-Onset Seizures in Adult Subjects With Drug-Resistant Epilepsy
Brief Title: A Study to Test the Efficacy and Safety of Padsevonil as Treatment of Focal-onset Seizures in Adult Subjects With Drug-resistant Epilepsy
Acronym: DUET
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Based on available data, UCB has decided to stop development of padsevonil as adjunctive treatment of focal-onset seizure
Sponsor: UCB Biopharma SRL (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EP0092; 2018-002303-33 (EudraCT Number)
Record Dates: First submitted 2018-11-09; First posted 2018-11-14 (Actual); Results first posted 2021-10-25 (Actual); Last update posted 2022-12-21 (Actual); Status verified 2022-12

CONDITIONS: Drug-Resistant Epilepsy; Focal-Onset Seizures
Keywords: Epilepsy; Padsevonil
MeSH Terms: conditions — Drug Resistant Epilepsy; Seizures; Epilepsy | interventions — padsevonil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Padsevonil dosing regimen 1 (Experimental): Subjects will be randomized to receive a combination of tablets of padsevonil and placebo (as appropriate) to maintain the blinding.
  Interventions: Drug: Padsevonil; Drug: Placebo
- Padsevonil dosing regimen 2 (Experimental): Subjects will be randomized to receive a combination of tablets of padsevonil and placebo (as appropriate) to maintain the blinding.
  Interventions: Drug: Padsevonil; Drug: Placebo
- Padsevonil dosing regimen 3 (Experimental): Subjects will be randomized to receive a combination of tablets of padsevonil and placebo (as appropriate) to maintain the blinding.
  Interventions: Drug: Padsevonil; Drug: Placebo
- Placebo (Placebo Comparator): Subjects randomized to the placebo group will receive a combination of several placebo tablets to maintain the blinding.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Padsevonil — Padsevonil in different dosages.
  Arms: Padsevonil dosing regimen 1; Padsevonil dosing regimen 2; Padsevonil dosing regimen 3
Drug: Placebo — Placebo will be provided matching padsevonil.

SUMMARY:
The purpose of the study is to evaluate the efficacy, safety and tolerability of the 3 selected dose regimens of padsevonil (PSL) administered concomitantly with up to 3 anti-epileptic drugs (AEDs) compared with placebo for treatment of observable focal-onset seizures in subjects with drug-resistant epilepsy.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of focal epilepsy per 1989 International League Against Epilepsy (ILAE) criteria at least 3 years before study entry
* Subject has failed to achieve seizure control with >=4 tolerated and appropriately chosen prior antiepileptic drugs (AED), including past and ongoing treatment, that were individually optimized for adequate dose and duration. Prior discontinued AED treatment would need to be assessed by the Investigator considering the patient medical records and patient and/or caregiver interview. 'Prior AED' is defined as all past and ongoing AED treatments with a start date before the Screening Visit (Visit 1)
* Average of >= 4 spontaneous and observable focal seizures (type IA1 (i.e. focal aware), IB (i.e. focal impaired awareness), IC (i.e. focal to bilateral tonic-clonic)) per month
* Current treatment with an individually optimized and stable dose of at least 1 and up to 3 AEDs for the 8 weeks prior to the Screening Visit with or without additional Vagus Nerve Stimulation (VNS) or other neurostimulation treatments

Exclusion Criteria:

* Subject has a history of or signs of generalized or combined generalized and focal epilepsy
* Cluster seizures which are uncountable in the previous 8 weeks before study entry and during 4 weeks prospective baseline
* Current treatment with carbamazepine, phenytoin, primidone, phenobarbital
* Current treatment/ use of (non-AED) prescription, nonprescription, dietary (eg, grapefruit or passion fruit), or herbal products that are potent inducers or inhibitors of the CYP3A4 or 2C19 pathway for 2 weeks (or 5 half-lives, whichever is longer) prior to the Baseline Visit
* Subjects taking sensitive substrates of CYP2C19 for 2 weeks (or 5 half-lives, whichever is longer) prior to the Baseline Visit
* Subject has been taking vigabatrin less than 2 years at study entry
* Subject has been taking felbamate for less than 12 months
* Subject taking retigabine for less than 4 years
* Current treatment with benzodiazepines (i.e. GABA-A-ergic drugs like zolpidem, zaleplon, or zopiclone, excluding GABA-A-ergic AEDs) <3 times per week for emergencies
* Subject has a current medical condition that occurred within the last 12 months which, in the opinion of the investigator, could compromise his/her safety or ability to participate in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 232 (Actual)
Dates: Start 2019-03-06 (Actual); Primary Completion 2020-09-28 (Actual); Study Completion 2020-09-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Cares, Study Director — 001 844 599 2273 (UCB)
Locations (141):
- United States (32):
  - Ep0092 839, Chandler, Arizona
  - Ep0092 881, Tucson, Arizona
  - Ep0092 633, Carlsbad, California
  - Ep0092 629, Orange, California
  - Ep0092 845, Washington D.C., District of Columbia
  - Ep0092 892, Bradenton, Florida
  - Ep0092 640, Hialeah, Florida
  - Ep0092 641, Jacksonville, Florida
  - Ep0092 823, Orlando, Florida
  - Ep0092 803, Honolulu, Hawaii
  - Ep0092 637, Urbana, Illinois
  - Ep0092 880, Anderson, Indiana
  - Ep0092 638, Fort Wayne, Indiana
  - Ep0092 630, Ames, Iowa
  - Ep0092 707, Lexington, Kentucky
  - Ep0092 822, Baltimore, Maryland
  - Ep0092 818, Bethesda, Maryland
  - Ep0092 889, Boston, Massachusetts
  - Ep0092 645, Golden Valley, Minnesota
  - Ep0092 644, Minneapolis, Minnesota
  - Ep0092 878, Brooklyn, New York
  - Ep0092 876, New York, New York
  - Ep0092 893, Syracuse, New York
  - Ep0092 895, The Bronx, New York
  - Ep0092 890, Chapel Hill, North Carolina
  - Ep0092 884, Charlotte, North Carolina
  - Ep0092 642, Columbus, Ohio
  - Ep0092 647, Oklahoma City, Oklahoma
  - Ep0092 882, Portland, Oregon
  - Ep0092 802, Philadelphia, Pennsylvania
  - Ep0092 829, Charlottesville, Virginia
  - Ep0092 639, Renton, Washington
- Australia (5):
  - Ep0092 855, Box Hill
  - Ep0092 861, Camperdown
  - Ep0092 850, Fitzroy
  - Ep0092 853, Heidelberg
  - Ep0092 852, Melbourne
- Belgium (2):
  - Ep0092 109, Brussels
  - Ep0092 107, Ottignies
- Bosnia and Herzegovina (4):
  - Ep0092 080, Bihać
  - Ep0092 077, Mostar
  - Ep0092 075, Sarajevo
  - Ep0092 082, Tuzla
- Bulgaria (4):
  - Ep0092 150, Blagoevgrad
  - Ep0092 151, Pleven
  - Ep0092 156, Pleven
  - Ep0092 154, Sofia
- Croatia (4):
  - Ep0092 125, Zagreb
  - Ep0092 126, Zagreb
  - Ep0092 127, Zagreb
  - Ep0092 128, Zagreb
- Czechia (4):
  - Ep0092 254, Brno
  - Ep0092 258, Ostrava
  - Ep0092 250, Prague
  - Ep0092 251, Prague
- Denmark (2):
  - Ep0092 016, Aarhus
  - Ep0092 015, Odense
- Estonia (3):
  - Ep0092 276, Tallinn
  - Ep0092 277, Tallinn
  - Ep0092 275, Tartu
- Ep0092 027, Tampere, Finland
- France (3):
  - Ep0092 312, Lyon
  - Ep0092 310, Paris
  - Ep0092 301, Strasbourg
- Germany (7):
  - Ep0092 365, Berlin
  - Ep0092 362, Bernau
  - Ep0092 363, Bielefeld
  - Ep0092 350, Frankfurt
  - Ep0092 368, Jena
  - Ep0092 357, Leipzig
  - Ep0092 376, Regensburg
- Greece (4):
  - Ep0092 425, Ioannina
  - Ep0092 426, Thessaloniki
  - Ep0092 427, Thessaloniki
  - Ep0092 428, Thessaloniki
- Hungary (3):
  - Ep0092 403, Budapest
  - Ep0092 405, Debrecen
  - Ep0092 404, Pécs
- Ireland (2):
  - Ep0092 035, Cork
  - Ep0092 036, Dublin
- Ep0092 452, Milan, Italy
- Japan (20):
  - Ep0092 526, Asahikawa
  - Ep0092 501, Asaka
  - Ep0092 521, Bunkyō City
  - Ep0092 525, Bunkyō City
  - Ep0092 504, Hamamatsu
  - Ep0092 505, Hiroshima
  - Ep0092 513, Hōfu
  - Ep0092 507, Itami
  - Ep0092 531, Izumi
  - Ep0092 539, Kumamoto
  - Ep0092 533, Kure
  - Ep0092 514, Kyoto
  - Ep0092 512, Nagakute
  - Ep0092 522, Ōmura
  - Ep0092 530, Ōsaka-sayama
  - Ep0092 515, Saitama
  - Ep0092 508, Sapporo
  - Ep0092 527, Shinagawa-Ku
  - Ep0092 509, Shizuoka
  - Ep0092 529, Yonago
- Ep0092 775, Sandvika, Norway
- Poland (12):
  - Ep0092 605, Katowice
  - Ep0092 616, Katowice
  - Ep0092 603, Krakow
  - Ep0092 614, Krakow
  - Ep0092 612, Lodz
  - Ep0092 610, Lublin
  - Ep0092 620, Lublin
  - Ep0092 606, Nowa Sól
  - Ep0092 611, Warsaw
  - Ep0092 615, Wroclaw
  - Ep0092 619, Zamość
  - Ep0092 618, Zgierz
- Portugal (2):
  - Ep0092 952, Aveiro
  - Ep0092 950, Matosinhos Municipality
- Romania (3):
  - Ep0092 925, Bucharest
  - Ep0092 926, Bucharest
  - Ep0092 927, Târgu Mureş
- Serbia (2):
  - Ep0092 327, Belgrade
  - Ep0092 325, Novi Sad
- Ep0092 004, Bardejov, Slovakia
- Spain (7):
  - Ep0092 662, Alicante
  - Ep0092 651, Barcelona
  - Ep0092 652, Barcelona
  - Ep0092 658, Barcelona
  - Ep0092 674, Madrid
  - Ep0092 657, Valencia
  - Ep0092 676, Zaragoza
- Sweden (2):
  - Ep0092 576, Gothenburg
  - Ep0092 575, Linköping
- Ep0092 053, Zurich, Switzerland
- Turkey (Türkiye) (6):
  - Ep0092 913, Ankara
  - Ep0092 915, Antalya
  - Ep0092 900, Istanbul
  - Ep0092 906, Istanbul
  - Ep0092 909, Istanbul
  - Ep0092 908, Trabzon
- United Kingdom (3):
  - Ep0092 766, Brighton
  - Ep0092 750, Manchester
  - Ep0092 764, Swansea

IPD SHARING:
Plan to Share IPD: Yes
Data from this trial may be requested by qualified researchers six months after product approval in the US and/or Europe, or global development is discontinued, and 18 months after trial completion. Investigators may request access to anonymized individual patient-level data and redacted trial documents which may include: analysis-ready datasets, study protocol, annotated case report form, statistical analysis plan, dataset specifications, and clinical study report. Prior to use of the data, proposals need to be approved by an independent review panel at www.Vivli.org and a signed data sharing agreement will need to be executed. All documents are available in English only, for a prespecified time, typically 12 months, on a password protected portal. This plan may change if the risk of re-identifying trial participants is determined to be too high after the trial is completed; in this case and to protect participants, individual patient-level data would not be made available.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data from this trial may be requested by qualified researchers six months after product approval in the US and/or Europe or global development is discontinued, and 18 months after trial completion.
Access Criteria: Qualified researchers may request access to anonymized IPD and redacted study documents which may include: raw datasets, analysis-ready datasets, study protocol, blank case report form, annotated case report form, statistical analysis plan, dataset specifications, and clinical study report. Prior to use of the data, proposals need to be approved by an independent review panel at www.Vivli.org and a signed data sharing agreement will need to be executed. All documents are available in English only, for a pre-specified time, typically 12 months, on a password protected portal.
URL: http://www.Vivli.org

REFERENCES:
- [Result] Rademacher M, Toledo M, Van Paesschen W, Liow KK, Milanov IG, Esch ML, Wang N, MacPherson M, Byrnes WJ, Minh TDC, Webster E, Werhahn KJ. Efficacy and safety of adjunctive padsevonil in adults with drug-resistant focal epilepsy: Results from two double-blind, randomized, placebo-controlled trials. Epilepsia Open. 2022 Dec;7(4):758-770. doi: 10.1002/epi4.12656. Epub 2022 Oct 22. PMID 36176044

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study started to enroll participants in March 2019 and concluded in September 2020.
Pre-assignment Details: The study included: a 4-week Baseline Period, a 16-week Treatment Period, a 4-week Taper Period (for participants who discontinued or choose not to enroll in the open-label extension study) and a Safety Follow-up Period. Participants continuing to the OLE study had a 3-week Conversion Period.
  The Participant Flow refers to the Randomized Set.
Groups:
- Placebo: Participants randomized to the placebo group received 5-6 placebo tablets to maintain the blinding, twice daily (bid) up to Week 19.
- Padsevonil 100 mg BID: Participants were randomized to receive a combination of tablets of padsevonil 100 mg and placebo (as appropriate) to maintain the blinding, bid up to Week 19.
- Padsevonil 200 mg BID: Participants were randomized to receive a combination of tablets of padsevonil 200 mg and placebo (as appropriate) to maintain the blinding, bid up to Week 19.
- Padsevonil 400 mg BID: Participants were randomized to receive a combination of tablets of padsevonil 400 mg and placebo (as appropriate) to maintain the blinding, bid up to Week 19
Period: Treatment Period: Wk0-16
Arm/Group | Placebo | Padsevonil 100 mg BID | Padsevonil 200 mg BID | Padsevonil 400 mg BID
Started | 56 | 60 | 57 | 59
Completed Titration and Stabilization | 54 | 58 | 51 | 54
Completed Maintenance Period | 46 | 44 | 44 | 36
Completed | 46 | 44 | 44 | 36
Not Completed | 10 | 16 | 13 | 23
Not completed — Adverse Event | 2 | 6 | 6 | 12
Not completed — Lack of Efficacy | 0 | 1 | 0 | 3
Not completed — Protocol Violation | 0 | 0 | 1 | 0
Not completed — Consent Withdrawn | 1 | 3 | 1 | 1
Not completed — Program Termination | 3 | 0 | 1 | 1
Not completed — Sponsor Closed Study- Subject Was Discontinued | 1 | 0 | 0 | 0
Not completed — Sponsors Decision | 3 | 2 | 1 | 3
Not completed — Promotor Decision | 0 | 1 | 0 | 0
Not completed — Per Sponsor Study Closed | 0 | 1 | 0 | 0
Not completed — Premature Program Termination | 0 | 1 | 0 | 0
Not completed — Trial Closed By Sponsor | 0 | 1 | 0 | 0
Not completed — Study Early Closure | 0 | 0 | 1 | 0
Not completed — Premature Study Termination By Sponsor | 0 | 0 | 1 | 0
Not completed — Premature Closure Of The Study | 0 | 0 | 1 | 0
Not completed — Study Has Been Cancelled By The Sponsor | 0 | 0 | 0 | 1
Not completed — Due To Sponsor Instruction | 0 | 0 | 0 | 1
Not completed — Trial Was Closed By Sponsor | 0 | 0 | 0 | 1
Period: Post-Treatment Period: Wk16-23
Arm/Group | Placebo | Padsevonil 100 mg BID | Padsevonil 200 mg BID | Padsevonil 400 mg BID
Started | 46 | 44 | 44 | 36
Started Conversion Period | 33 | 31 | 29 | 28
Completed Conversion Period | 33 | 31 | 29 | 28
Started Taper and Safety Follow-up | 19 | 18 | 21 | 13
Completed Taper and Safety Follow-up | 15 | 16 | 18 | 12
Enrolled in EP0093 | 27 | 26 | 23 | 23
Completed | 42 | 42 | 41 | 35
Not Completed | 4 | 2 | 3 | 1
Not completed — Adverse Event | 3 | 0 | 0 | 0
Not completed — Consent Withdrawn | 0 | 0 | 0 | 1
Not completed — Sponsor Decision To Terminate The Study | 1 | 0 | 0 | 0
Not completed — Sponsor's Decision | 0 | 1 | 0 | 0
Not completed — Sponsor Closed Study- Subject Was Discontinued | 0 | 1 | 0 | 0
Not completed — Sponsor Decision + Subject Refusal | 0 | 0 | 1 | 0
Not completed — Early Study Closure | 0 | 0 | 1 | 0
Not completed — Trial Closed By Sponsor Decision | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Baseline Characteristics refer to the Randomized Set (RS) consisted of all participants randomized into the study.
Arm/Group | Placebo | Padsevonil 100 mg BID | Padsevonil 200 mg BID | Padsevonil 400 mg BID | Total Title
Number analyzed (Participants) | 56 | 60 | 57 | 59 | 232
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1 | 0 | 4 | 0 | 5
  Between 18 and 65 years | 52 | 57 | 48 | 56 | 213
  >=65 years | 3 | 3 | 5 | 3 | 14
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.9 (13.6) | 40.7 (13.0) | 39.5 (14.3) | 39.7 (13.6) | 40.4 (13.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34 | 34 | 29 | 34 | 131
  Male | 22 | 26 | 28 | 25 | 101
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 0 | 0 | 1
  Asian | 5 | 5 | 7 | 7 | 24
  Black | 0 | 1 | 1 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 2 | 0 | 0 | 2
  White | 49 | 50 | 49 | 51 | 199
  Other/mixed | 1 | 2 | 0 | 0 | 3

OUTCOME MEASURES:

1. Primary Outcome: Change in Log-transformed Observable Focal-onset Seizure Frequency From Baseline Over the 12-week Maintenance Period
Description: During the study, participants kept diaries to record daily seizure activity. Seizure frequency refers to 28-day adjusted frequency. Seizure frequency was based on investigator assessment of participants' reports of daily seizure type and frequency. Observable focal-onset seizures refer to Type IA1, IB, and IC (ILAE Classification of Epileptic Seizures, 1981). Based on ANCOVA on change in log-transformed seizure frequency from Baseline, with treatment group as the main factor, Baseline log-transformed seizure frequency as a continuous covariate, Baseline SV2A use (Yes or No) and Region (Europe, non-Europe) as categorical factors.
Time Frame: From Baseline over the 12 Week Maintenance Period (up to Week 16)
Population: The Full Analysis Set (FAS) consisted of all study participants in the RS who were administered at least 1 dose or a partial dose of IMP and had Baseline and at least 1 post-Baseline seizure frequency data during the 16-week Treatment Period. Here, number of participants were included who were evaluable for the assessment.
Measure: Least Squares Mean (95% Confidence Interval); unit: log e seizures per 28 days
Groups:
- Placebo (FAS): Participants randomized to the placebo group received 5-6 placebo tablets to maintain the blinding, bid up to Week 19. Participants formed the Full Analysis Set (FAS).
- Padsevonil 100 mg BID (FAS): Participants were randomized to receive a combination of tablets of padsevonil 100 mg and placebo (as appropriate) to maintain the blinding, bid up to Week 19. Participants formed the FAS.
- Padsevonil 200 mg BID (FAS): Participants were randomized to receive a combination of tablets of padsevonil 200 mg and placebo (as appropriate) to maintain the blinding, bid up to Week 19. Participants formed the FAS.
- Padsevonil 400 mg BID (FAS): Participants were randomized to receive a combination of tablets of padsevonil 400 mg and placebo (as appropriate) to maintain the blinding, bid up to Week 19. Participants formed the FAS.
Arm/Group | Placebo (FAS) | Padsevonil 100 mg BID (FAS) | Padsevonil 200 mg BID (FAS) | Padsevonil 400 mg BID (FAS)
Number analyzed (Participants) | 54 | 59 | 56 | 56
log e seizures per 28 days | -0.41 [-0.6133 to -0.2025] | -0.35 [-0.54906 to -0.15705] | -0.47 [-0.67559 to -0.27382] | -0.47 [-0.67267 to -0.27361]
Statistical Analysis 1: Comparison: Placebo (FAS) vs Padsevonil 100 mg BID (FAS); Percent reduction over placebo was calculated as 100*(1-exp(diff)), where diff was the model estimate of the log ratio between each PSL group and placebo group; Test type: Superiority; p = 0.687, ANCOVA — Adjusted p-values are from the Hochberg step-up procedure within SAS® Proc Multtest to control Type I error; Percent reduction = -5.6, 95% CI 2-sided [-38.1 to 19.2]
Statistical Analysis 2: Comparison: Placebo (FAS) vs Padsevonil 200 mg BID (FAS); [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.687, ANCOVA — Adjusted p-values were from the Hochberg step-up procedure within SAS® Proc Multtest to control Type I error; Percent reduction = 6.5, 95% CI 2-sided [-22.7 to 28.7]
Statistical Analysis 3: Comparison: Placebo (FAS) vs Padsevonil 400 mg BID (FAS); [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.687, ANCOVA — Adjusted p-values were from the Hochberg step-up procedure within SAS® Proc Multtest to control Type I error; Percent reduction = 6.3, 95% CI 2-sided [-22.9 to 28.6]

2. Primary Outcome: Percentage of Participants With Treatment-Emergent Adverse Events (TEAEs)
Description: An Adverse Event is any untoward medical occurrence in a patient or clinical investigation subject administered a pharmaceutical product that does not necessarily have a causal relationship with this treatment. A TEAE was defined as any event not present before the initiation of the first dose of study treatment or any unresolved event already present before initiation of the first dose that worsened in intensity following exposure to the treatment.
Time Frame: From Baseline until Safety Follow-Up (up to Week 23)
Population: The Safety Set consisted of all study participants who were administered at least 1 dose or a partial dose of IMP.
Measure: Number; unit: percentage of participants
Groups:
- Placebo (SS): Participants randomized to the placebo group received 5-6 placebo tablets to maintain the blinding, bid up to Week 19. Participants formed the Safety Set (SS).
- Padsevonil 100 mg BID (SS): Participants were randomized to receive a combination of tablets of padsevonil 100 mg and placebo (as appropriate) to maintain the blinding, bid up to Week 19. Participants formed the SS.
- Padsevonil 200 mg BID (SS): Participants were randomized to receive a combination of tablets of padsevonil 200 mg and placebo (as appropriate) to maintain the blinding, bid up to Week 19. Participants formed the SS.
- Padsevonil 400 mg BID (SS): Participants were randomized to receive a combination of tablets of padsevonil 400 mg and placebo (as appropriate) to maintain the blinding, bid up to Week 19. Participants formed the SS.
Arm/Group | Placebo (SS) | Padsevonil 100 mg BID (SS) | Padsevonil 200 mg BID (SS) | Padsevonil 400 mg BID (SS)
Number analyzed (Participants) | 55 | 60 | 57 | 59
percentage of participants | 69.1 | 83.3 | 78.9 | 84.7

3. Primary Outcome: Percentage of Participants With Treatment-Emergent Adverse Events (TEAEs) Leading to Study Withdrawal
Description: as for outcome 2
Time Frame: From Baseline until Safety Follow-Up (up to Week 23)
Population: The Safety Set consisted of all study participants who were administered at least 1 dose or a partial dose of IMP.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo (SS) | Padsevonil 100 mg BID (SS) | Padsevonil 200 mg BID (SS) | Padsevonil 400 mg BID (SS)
Number analyzed (Participants) | 55 | 60 | 57 | 59
percentage of participants | 7.3 | 10.0 | 10.5 | 20.3

4. Primary Outcome: Percentage of Participants With Treatment-Emergent Serious Adverse Events (SAEs)
Description: A Serious Adverse Event (SAE) is any untoward medical occurrence that at any dose: Results in death, is life-threatening, requires in patient hospitalization or prolongation of existing hospitalization, is a congenital anomaly or birth defect, is as infection that requires treatment parenteral antibiotics, other important medical events which based on medical or scientific judgement may jeopardize the patients, or may require medical or surgical intervention to prevent any of the above. A TEAE was defined as any event not present before the initiation of the first dose of study treatment or any unresolved event already present before initiation of the first dose that worsened in intensity following exposure to the treatment.
Time Frame: From Baseline until Safety Follow-Up (up to Week 23)
Population: The Safety Set consisted of all study participants who were administered at least 1 dose or a partial dose of IMP.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo (SS) | Padsevonil 100 mg BID (SS) | Padsevonil 200 mg BID (SS) | Padsevonil 400 mg BID (SS)
Number analyzed (Participants) | 55 | 60 | 57 | 59
percentage of participants | 9.1 | 3.3 | 1.8 | 10.2

5. Secondary Outcome: 75% Responder Rate From Baseline Over the 12-week Maintenance Period
Description: The 75 % responder rate, where a responder was a participant experiencing a ≥75 % reduction in observable focal-onset seizure frequency from Baseline, over the 12-Week Maintenance Period.
Time Frame: From Baseline over the 12 Week Maintenance Period (up to Week 16)
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Placebo (FAS) | Padsevonil 100 mg BID (FAS) | Padsevonil 200 mg BID (FAS) | Padsevonil 400 mg BID (FAS)
Number analyzed (Participants) | 54 | 59 | 56 | 56
percentage of participants | 13.0 | 15.3 | 12.5 | 14.3
Statistical Analysis 1: Comparison: Placebo (FAS) vs Padsevonil 100 mg BID (FAS); PSL dose/Placebo calculated using logistic regression with categorical factors for treatment group (each PSL dose group referenced to the placebo group), Region (Europe, non-Europe), Baseline SV2A use (Yes, No) and log-transformed Baseline seizure frequency as a continuous covariate; Test type: Superiority; p = 0.803, Regression, Logistic — Nominal p-values were not adjusted for multiplicity; Odds Ratio (OR) = 1.15, 95% CI 2-sided [0.39 to 3.38]
Statistical Analysis 2: Comparison: Placebo (FAS) vs Padsevonil 200 mg BID (FAS); [analysis description as in outcome 5, analysis 1]; Test type: Superiority; p = 0.772, Regression, Logistic — Nominal p-values were not adjusted for multiplicity; Odds Ratio (OR) = 0.84, 95% CI 2-sided [0.27 to 2.65]
Statistical Analysis 3: Comparison: Placebo (FAS) vs Padsevonil 400 mg BID (FAS); [analysis description as in outcome 5, analysis 1]; Test type: Superiority; p = 0.989, Regression, Logistic — Nominal p-values were not adjusted for multiplicity; Odds Ratio (OR) = 1.01, 95% CI 2-sided [0.33 to 3.08]

6. Secondary Outcome: 50% Responder Rate From Baseline Over the 12-week Maintenance Period
Description: The 50% responder rate, where a responder was a participant experiencing a ≥50% reduction in observable focal-onset seizure frequency from Baseline, over the 12-week Maintenance Period.
Time Frame: From Baseline over the 12 Week Maintenance Period (up to Week 16)
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Placebo (FAS) | Padsevonil 100 mg BID (FAS) | Padsevonil 200 mg BID (FAS) | Padsevonil 400 mg BID (FAS)
Number analyzed (Participants) | 54 | 59 | 56 | 56
percentage of participants | 27.8 | 35.6 | 33.9 | 42.9
Statistical Analysis 1: Comparison: Placebo (FAS) vs Padsevonil 100 mg BID (FAS); [analysis description as in outcome 5, analysis 1]; Test type: Superiority; p = 0.425, Regression, Logistic — Nominal p-values were not adjusted for multiplicity; Odds Ratio (OR) = 1.40, 95% CI 2-sided [0.61 to 3.18]
Statistical Analysis 2: Comparison: Placebo (FAS) vs Padsevonil 200 mg BID (FAS); [analysis description as in outcome 5, analysis 1]; Test type: Superiority; p = 0.625, Regression, Logistic — Nominal p-values were not adjusted for multiplicity; Odds Ratio (OR) = 1.23, 95% CI 2-sided [0.53 to 2.85]
Statistical Analysis 3: Comparison: Placebo (FAS) vs Padsevonil 400 mg BID (FAS); [analysis description as in outcome 5, analysis 1]; Test type: Superiority; p = 0.125, Regression, Logistic — Nominal p-values were not adjusted for multiplicity; Odds Ratio (OR) = 1.90, 95% CI 2-sided [0.84 to 4.34]

7. Secondary Outcome: Percent Change in Observable Focal-onset Seizure Frequency From Baseline Over the 12-week Maintenance Period
Description: During the study, participants kept diaries to record daily seizure activity. The percentage of participants who experienced a 50 % or greater reduction in seizure frequency per 28 days relative to Baseline (responders) were assessed.
Time Frame: From Baseline over the 12 Week Maintenance Period (up to Week 16)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo (FAS) | Padsevonil 100 mg BID (FAS) | Padsevonil 200 mg BID (FAS) | Padsevonil 400 mg BID (FAS)
Number analyzed (Participants) | 54 | 59 | 56 | 56
percent change | 22.34 (44.56) | 11.72 (81.52) | 30.29 (39.58) | 22.41 (62.80)
Statistical Analysis 1: Comparison: Placebo (FAS) vs Padsevonil 100 mg BID (FAS); Dose group comparisons to Placebo p-value are based on the Wilcoxon-Mann-Whitney test. Hodges Lehmann nonparametric effect estimates and corresponding two-sided 95% asymptotic confidence intervals are provided for the effect difference between each PSL dose and placebo; Test type: Superiority; p = 0.737, Wilcoxon (Mann-Whitney) — Nominal p-values were not adjusted for multiplicity; Median Difference (Final Values) = 3.25, 95% CI 2-sided [-17.08 to 20.36]
Statistical Analysis 2: Comparison: Placebo (FAS) vs Padsevonil 200 mg BID (FAS); [analysis description as in outcome 7, analysis 1]; Test type: Superiority; p = 0.458, Wilcoxon (Mann-Whitney) — Nominal p-values were not adjusted for multiplicity; Median Difference (Net) = 6.17, 95% CI 2-sided [-10.00 to 21.91]
Statistical Analysis 3: Comparison: Placebo (FAS) vs Padsevonil 400 mg BID (FAS); [analysis description as in outcome 7, analysis 1]; Test type: Superiority; p = 0.341, Wilcoxon (Mann-Whitney) — Nominal p-values were not adjusted for multiplicity; Median Difference (Net) = 9.31, 95% CI 2-sided [-10.92 to 28.21]

ADVERSE EVENTS:
Time Frame: TEAEs were collected from Baseline until Safety Follow-Up (up to Week 23)
Description: TEAEs counts are for the number of study participants who entered the respective study period regardless of whether or not they completed the previous period. This is the reason for the difference in number of participants in Taper and SFU period in adverse events section and participant flow.
Groups:
- Placebo Treatment Period (SS): Participants randomized to the placebo group received 5-6 placebo tablets to maintain the blinding, bid up to Week 19. Participants formed the Safety Set (SS).
- Padsevonil 100 mg BID Treatment Period (SS): Participants were randomized to receive a combination of tablets of padsevonil 100 mg and placebo (as appropriate) to maintain the blinding, bid up to Week 19. Participants formed the SS.
- Padsevonil 200 mg BID Treatment Period (SS): Participants were randomized to receive a combination of tablets of padsevonil 200 mg and placebo (as appropriate) to maintain the blinding, bid up to Week 19. Participants formed the SS.
- Padsevonil 400 mg BID Treatment Period (SS): Participants were randomized to receive a combination of tablets of padsevonil 400 mg and placebo (as appropriate) to maintain the blinding, bid up to Week 19. Participants formed the SS.
- Placebo Conversion Period (SS): A 3-Week Conversion Period was required for study participants who chose to enroll in the open-label extension (OLE) study at the end of the 12-Week Maintenance Period. Participants initially randomized to placebo progressively received padsevonil in a blinded way to reach the entry dose of 400 mg/day for the OLE. Participants formed the Safety Set (SS).
- Padsevonil 100 mg BID Conversion Period (SS): A 3-Week Conversion Period was required for study participants who chose to enroll in the OLE study at the end of the 12-Week Maintenance Period. The dose for participants initially randomized to padsevonil 100 mg bid was gradually adapted (increased or decreased) in a blinded way to reach the entry dose of 400 mg/day for the OLE. Participants formed the SS.
- Padsevonil 200 mg BID Conversion Period (SS): A 3-Week Conversion Period was required for study participants who chose to enroll in the OLE study at the end of the 12-Week Maintenance Period. The dose for participants initially randomized to padsevonil 200 mg bid was gradually adapted (increased or decreased) in a blinded way to reach the entry dose of 400 mg/day for the OLE. Participants formed the SS.
- Padsevonil 400 mg BID Conversion Period (SS): A 3-Week Conversion Period was required for study participants who chose to enroll in the OLE study at the end of the 12-Week Maintenance Period. The dose for participants initially randomized to padsevonil 400 mg bid was gradually adapted (increased or decreased) in a blinded way to reach the entry dose of 400 mg/day for the OLE. Participants formed the SS.
- Placebo Taper and SFU Period (SS): A 4-Week Taper Period was required for participants who chose not to enroll in the OLE study or who discontinued prior to the end of the 12-Week Maintenance Period. Participants initially randomized to placebo group received 5-6 placebo tablets to maintain the blinding and have been gradually tapered off the IMP over a 3-week period followed by 1-week drug-free period. Afterwards, participants had a Safety Follow-Up visit 30 days after the last IMP intake. Participants formed the Safety Set (SS).
- Padsevonil 100 mg BID Taper and SFU Period (SS): A 4-Week Taper Period was required for participants who chose not to enroll in the OLE study or who discontinued prior to the end of the 12-Week Maintenance Period. Participants initially randomized to padsevonil 100 mg bid have been gradually tapered off the IMP over a 3-week period followed by 1-week drug-free period. Afterwards, participants had a Safety Follow-Up visit 30 days after the last IMP intake. Participants formed the SS.
- Padsevonil 200 mg BID Taper and SFU Period (SS): A 4-Week Taper Period was required for participants who chose not to enroll in the OLE study or who discontinued prior to the end of the 12-Week Maintenance Period. Participants initially randomized to padsevonil 200 mg bid have been gradually tapered off the IMP over a 3-week period followed by 1-week drug-free period. Afterwards, participants had a Safety Follow-Up visit 30 days after the last IMP intake. Participants formed the SS.
- Padsevonil 400 mg BID Taper and SFU Period (SS): A 4-Week Taper Period was required for participants who chose not to enroll in the OLE study or who discontinued prior to the end of the 12-Week Maintenance Period. Participants initially randomized to padsevonil 400 mg bid have been gradually tapered off the IMP over a 3-week period followed by 1-week drug-free period. Afterwards, participants had a Safety Follow-Up visit 30 days after the last IMP intake. Participants formed the SS.
Arm/Group | Placebo Treatment Period (SS) | Padsevonil 100 mg BID Treatment Period (SS) | Padsevonil 200 mg BID Treatment Period (SS) | Padsevonil 400 mg BID Treatment Period (SS) | Placebo Conversion Period (SS) | Padsevonil 100 mg BID Conversion Period (SS) | Padsevonil 200 mg BID Conversion Period (SS) | Padsevonil 400 mg BID Conversion Period (SS) | Placebo Taper and SFU Period (SS) | Padsevonil 100 mg BID Taper and SFU Period (SS) | Padsevonil 200 mg BID Taper and SFU Period (SS) | Padsevonil 400 mg BID Taper and SFU Period (SS)
All-Cause Mortality (participants affected / at risk) | 0/55 | 0/60 | 0/57 | 0/59 | 0/33 | 0/31 | 0/29 | 0/28 | 0/27 | 0/30 | 0/31 | 0/32
Serious Adverse Events (participants affected / at risk) | 3/55 | 0/60 | 1/57 | 5/59 | 1/33 | 0/31 | 0/29 | 0/28 | 1/27 | 2/30 | 0/31 | 1/32
Other Adverse Events (participants affected / at risk) | 25/55 | 37/60 | 40/57 | 41/59 | 7/33 | 0/31 | 1/29 | 1/28 | 2/27 | 6/30 | 4/31 | 2/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo Treatment Period (SS) (N=55) | Padsevonil 100 mg BID Treatment Period (SS) (N=60) | Padsevonil 200 mg BID Treatment Period (SS) (N=57) | Padsevonil 400 mg BID Treatment Period (SS) (N=59) | Placebo Conversion Period (SS) (N=33) | Padsevonil 100 mg BID Conversion Period (SS) (N=31) | Padsevonil 200 mg BID Conversion Period (SS) (N=29) | Padsevonil 400 mg BID Conversion Period (SS) (N=28) | Placebo Taper and SFU Period (SS) (N=27) | Padsevonil 100 mg BID Taper and SFU Period (SS) (N=30) | Padsevonil 200 mg BID Taper and SFU Period (SS) (N=31) | Padsevonil 400 mg BID Taper and SFU Period (SS) (N=32)
Radius fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin laceration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Wrist fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Epilepsy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Focal dyscognitive seizures (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Status epilepticus (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Aggression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Emotional disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abortion induced (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Placebo Treatment Period (SS) (N=55) | Padsevonil 100 mg BID Treatment Period (SS) (N=60) | Padsevonil 200 mg BID Treatment Period (SS) (N=57) | Padsevonil 400 mg BID Treatment Period (SS) (N=59) | Placebo Conversion Period (SS) (N=33) | Padsevonil 100 mg BID Conversion Period (SS) (N=31) | Padsevonil 200 mg BID Conversion Period (SS) (N=29) | Padsevonil 400 mg BID Conversion Period (SS) (N=28) | Placebo Taper and SFU Period (SS) (N=27) | Padsevonil 100 mg BID Taper and SFU Period (SS) (N=30) | Padsevonil 200 mg BID Taper and SFU Period (SS) (N=31) | Padsevonil 400 mg BID Taper and SFU Period (SS) (N=32)
Nausea (Gastrointestinal disorders) | 3 (5) | 1 (1) | 3 (4) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 3 (4) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 4 (4) | 5 (5) | 7 (7) | 14 (15) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Asthenia (General disorders) | 2 (2) | 6 (6) | 3 (4) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gait disturbance (General disorders) | 0 (0) | 2 (2) | 2 (3) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 4 (4) | 1 (1) | 4 (4) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 3 (4) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 3 (4) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 2 (2) | 10 (11) | 19 (22) | 20 (23) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 4 (5) | 14 (14) | 10 (13) | 18 (19) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 8 (13) | 10 (22) | 9 (16) | 5 (8) | 0 (0) | 0 (0) | 0/28 (0) | 0/27 (0) | 0 (0) | 4 (12) | 2 (2) | 1 (1)
Memory impairment (Nervous system disorders) | 1 (1) | 0 (0) | 3 (3) | 6 (6) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tremor (Nervous system disorders) | 1 (1) | 3 (5) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Disturbance in attention (Nervous system disorders) | 1 (1) | 1 (1) | 5 (5) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Balance disorder (Nervous system disorders) | 0 (0) | 1 (1) | 3 (3) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dysarthria (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 5 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 1 (1) | 0 (0) | 4 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1) | 5 (6) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Irritability (Psychiatric disorders) | 3 (3) | 4 (4) | 3 (3) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (2) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2020-01-21): https://cdn.clinicaltrials.gov/large-docs/40/NCT03739840/Prot_000.pdf
  • Statistical Analysis Plan (2020-08-18): https://cdn.clinicaltrials.gov/large-docs/40/NCT03739840/SAP_001.pdf